CLINICAL TRIAL: NCT06106568
Title: A Retrospective Observational Study to Investigate the Clinical Impact of EOB-MRI in the Diagnosis of Liver Metastasis of Pancreatic Cancer in Japan - A Real-World Study
Brief Title: An Observational Study to Learn More About the Impact of Gadoxetate Sodium-Enhanced Magnetic Resonance Imaging (EOB-MRI) When Used to Diagnose the Spread of Cancer From the Pancreas to the Liver in Japanese People Under Real-World Conditions
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22470
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Pancreatic Cancer; Liver Metastases; Gadoxetate Sodium-enhanced Magnetic Resonance Imaging
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- EOB-MRI: Adult patients with confirmed diagnosis of pancreatic cancer who had the prescription record of an active treatment preceding the pancreatic cancer diagnosis and with a record of EOB-MRI
  Interventions: Procedure: EOB-MRI
- non-EOB-MRI: Adult patients with confirmed diagnosis of pancreatic cancer who had the prescription record of an active treatment preceding the pancreatic cancer diagnosis and without a record of EOB-MBI
- EOB-MRI with surgery: Adult patients with confirmed diagnosis of pancreatic cancer who had the prescription record of an active treatment preceding the pancreatic cancer diagnosis and with a record of EOB-MRI and surgery
  Interventions: Procedure: EOB-MRI; Procedure: Surgery
- non-EOB-MRI with surgery: Adult patients with confirmed diagnosis of pancreatic cancer who had the prescription record of an active treatment preceding the pancreatic cancer diagnosis and without a record of EOB-MRI but with a record of surgery
  Interventions: Procedure: Surgery
- EOB-MRI without surgery: Adult patients with confirmed diagnosis of pancreatic cancer who had the prescription record of an active treatment preceding the pancreatic cancer diagnosis and with a record of EOB-MRI but without a record of surgery
  Interventions: Procedure: EOB-MRI
- non-EOB-MRI without surgery: Adult patients with confirmed diagnosis of pancreatic cancer who had the prescription record of an active treatment preceding the pancreatic cancer diagnosis and without a record of EOB-MRI or surgery
- EOB-MRI with an open-close laparotomy: Adult patients with confirmed diagnosis of pancreatic cancer who had the prescription record of an active treatment preceding the pancreatic cancer diagnosis and with a record of EOB-MRI and an open-close laparotomy
  Interventions: Procedure: EOB-MRI; Procedure: Open-close Laparotomy
- non-EOB-MRI with an open-close laparotomy: Adult patients with confirmed diagnosis of pancreatic cancer who had the prescription record of an active treatment preceding the pancreatic cancer diagnosis and without a record of EOB-MRI but with a record of an open-close laparotomy
  Interventions: Procedure: Open-close Laparotomy

INTERVENTIONS:
Procedure: EOB-MRI — Retrospective analysis for pancreatic cancer patients who had a record of EOB-MRI in the Medical Data Vision (MDV) database in Japan
  Groups: EOB-MRI; EOB-MRI with an open-close laparotomy; EOB-MRI with surgery; EOB-MRI without surgery
Procedure: Surgery — Retrospective analysis for pancreatic cancer patients who had a record of any surgery for the pancreatic cancer in the Medical Data Vision (MDV) database in Japan
  Groups: EOB-MRI with surgery; non-EOB-MRI with surgery
Procedure: Open-close Laparotomy — Retrospective analysis for pancreatic cancer patients who had a record of an open-close laparotomy in the Medical Data Vision (MDV) database in Japan
  Groups: EOB-MRI with an open-close laparotomy; non-EOB-MRI with an open-close laparotomy

SUMMARY:
This is an observational study in which data from people with cancer that has spread from the pancreas to the liver are collected and studied. These adults will include people who already received their usual treatment and who have had a certain type of imaging scan before the diagnosis of pancreatic cancer.

Metastatic pancreatic cancer is a cancer that starts in the pancreas, a gland that helps to digest food, and has spread to other parts of the body. Pancreatic cancer most commonly spreads to the liver (called liver metastasis). Gadoxetate sodium-enhanced magnetic resonance imaging (EOB-MRI) is a type of imaging technique that uses a specific dye called gadoxetate sodium to produce clearer images of the liver.

Participants with pancreatic cancer can be treated with surgery only if their cancer has not spread to other parts of the body. Therefore, it is important to find out if the cancer has spread to other parts of the body before performing surgery. To do this, different imaging scans such as exploratory laparoscopy and CE-CT are used. However, these tests have certain limitations, such as complicated procedures or, in some cases inaccurate results.

Some studies suggest that performing EOB-MRI along with a regular CT scan may improve the chances of finding out if pancreatic cancer has spread to the liver. This imaging technique is especially helpful in detecting smaller tumors that may be missed in other types of scan. However, more information is needed to better understand the impact of EOB-MRI in Japanese people under real-world conditions.

The main purpose of this study is to learn more about how using EOB-MRI helps in deciding the treatment options, how well the participants do, and how much does the use of medical care facilities costs.

The main information that researchers will collect in this study:

participant characteristics, including age, sex, whether they smoke or not, how well they can manage daily tasks, any other health problems they have, how advanced their cancer is, and if they have undergone laparoscopy

the length of time:

from the date of diagnosis of pancreatic cancer until a participant dies (called overall survival)

from the date of first treatment for pancreatic cancer until the cancer spreads of other organs

from the date of diagnosis of pancreatic cancer to starting the first treatment

from the date of first treatment for pancreatic cancer to starting the second treatment option

treatments that the participants have received, including anti-cancer drugs, radiation, and surgery

the number of hospital visits, use of healthcare facilities, and related costs.

The information in this study will be grouped based on the participants who had an EOB-MRI and those who had non EOB-MRI.

The data will come from the participants' information stored in a database called Medical Data Vision (MDV) in Japan. Data collected will be from January 2011 to October 2022.

Researchers will track individual patients' data for at least 1 year, until death, until there is no health record in the MDV for 2 months after treatment starts, or until the end of study.

In this study, only available data from health records are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients having at least one confirmed diagnosis of pancreatic cancer (identified by ICD-10 diagnosis code C25.x, without a suspicious diagnosis flag) during the patient selection period
* Patients having at least one active treatment record after the 1st confirmed diagnosis of pancreatic cancer
* Patients 18 years of age or older at the index date
* Patients having any recorded CE-CT or EOB-MRI or MRI without EOB record during the baseline period

  * EOB-MRI stands for enhanced liver MRI using gadoxetate sodium as the contrast agent. In this type of MRI, gadoxetate sodium is used as a contrast agent in the visualization of the liver tumor.
  * EOB-MRI group will include patients who underwent EOB-MRI during the baseline period.
  * Non-EOB-MRI group will include patients who underwent CE-CT or MRI with contrast agent other than the gadoxetate sodium during the baseline period.
  * MRI, CE-CT and contrast agents are identified by using the nine-digit Japanese receipt code specified in the separate code list

Exclusion Criteria:

* Patients with no confirmed diagnosis of pancreatic cancer (ICD-10 diagnosis code C25.x) in the below category of the disease name in the discharge summary until the 1st discharge date after the index date:

  * "ICD-10 code of disease name which input the most medical resources"
  * "ICD-10 name of disease behind hospitalization"
* Patients with no active treatment within 3 months (90 days) from the con-firmed pancreatic cancer diagnosis date
* Patients with no medical record in the MDV database within 1 month (30 days) from the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective observational study utilizing data extracted from a hospital-based administrative health insurance claims database provided by Medical Data Vision Co. Ltd (MDV, Tokyo, Japan). Eligible patients are adult patients with a confirmed diagnosis of pancreatic cancer (identified by International Classification of Diseases, 10th revision [ICD-10] code C25.x) during the overall study period (i.e., between 01 Jan 2011 and 31 Oct 2022) .
Sampling Method: Non-Probability Sample
Enrollment: 39624 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Descriptive summary of patient characteristics in EOB-MRI and non-EOB-MRI group | Up to 12 years
Descriptive summary of treatment pathways in EOB-MRI and non-EOB-MRI group | Up to 12 years
Descriptive summary of healthcare utilization patterns in EOB-MRI and non-EOB-MRI group | Up to 12 years
Descriptive summary of healthcare costs in EOB-MRI and non-EOB-MRI group | Up to 12 years

SECONDARY OUTCOMES:
Descriptive summary of patient characteristics in EOB-MRI and non-EOB-MRI group within the subgroups of interest | Up to 12 years
  Subgroups:
  * with a record of surgery
  * without a record of surgery
  * with a record of an open-close laparotomy
Descriptive summary of clinical outcomes in EOB-MRI and non-EOB-MRI group within the subgroups of interest | Up to 12 years
  Subgroups:
  * with a record of surgery
  * without a record of surgery
  * with a record of an open-close laparotomy
Descriptive summary of healthcare utilization pattern in EOB-MRI and non-EOB-MRI group within the subgroups of interest | Up to 12 years
  Subgroups:
  * with a record of surgery
  * without a record of surgery
  * with a record of an open-close laparotomy
Descriptive summary of healthcare costs in EOB-MRI and non-EOB-MRI group within the subgroups of interest | Up to 12 years
  Subgroups:
  * with a record of surgery
  * without a record of surgery
  * with a record of an open-close laparotomy
Comparison of overall survival (time from pancreatic cancer diagnosis date to death) (in days) between patients in the EOB-MRI and non-EOB-MRI groups within the subgroups of interest (surgery and non-surgery) | Up to 12 years
Comparison of time to diagnosis of new metastases from the index date (in days) between patients in the EOB-MRI and non-EOB-MRI groups within the subgroups of interest (surgery and non-surgery) | Up to 12 years
Comparison of time to first treatment pathway option from the pancreatic cancer diagnosis date (in days) between patients in the EOB-MRI and non-EOB-MRI groups within the subgroups of interest (surgery and non-surgery) | Up to 12 years
Comparison of time to second treatment pathway option from the index date (in days) between patients in the EOB-MRI and non-EOB-MRI groups within the subgroups of interest (surgery and non-surgery) | Up to 12 years
Descriptive summary of patient characteristics across three index-year groups | Up to 12 years
  The study period will be divided into index year groups defined as below:
  * Group 1: 2011-2012
  * Group 2: 2013-2018
  * Group 3: 2019-2021
Descriptive summary of clinical outcomes across three index-year groups | Up to 12 years
  The study period will be divided into index year groups defined as below:
  * Group 1: 2011-2012
  * Group 2: 2013-2018
  * Group 3: 2019-2021
Descriptive summary of treatment pathways across three index-year groups | Up to 12 years
  The study period will be divided into index year groups defined as below:
  * Group 1: 2011-2012
  * Group 2: 2013-2018
  * Group 3: 2019-2021
Descriptive summary of healthcare utilization pattern across three index-year groups | Up to 12 years
  The study period will be divided into index year groups defined as below:
  * Group 1: 2011-2012
  * Group 2: 2013-2018
  * Group 3: 2019-2021
Descriptive summary of healthcare costs across three index-year groups | Up to 12 years
  The study period will be divided into index year groups defined as below:
  * Group 1: 2011-2012
  * Group 2: 2013-2018
  * Group 3: 2019-2021
Descriptive summary of the likelihood of open-close laparotomy in patients with confirmed diagnosis of pancreatic cancer who is intended the surgical intervention between those in the EOB-MRI group and non-EOB-MRI group | Up to 12 years

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.